CLINICAL TRIAL: NCT00919984
Title: Phase II Clinical Trial of Intravenous Paclitaxel and Carboplatin Plus Intraperitoneal Paclitaxel as an Adjuvant Chemotherapy in Patients With Optimally Debulked Advanced Epithelial Ovarian Carcinoma
Brief Title: Efficacy Study of Additional Intraperitoneal Chemotherapy to Treat Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study stopped due to slow accrual.
Sponsor: Korea Cancer Center Hospital (Other)
Responsible Party: Principal Investigator, Sang-Young Ryu, Chair of Cerivcal/Ovarian Cancer Center, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCCH GY 3001
Record Dates: First submitted 2009-06-07; First posted 2009-06-12 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Ovarian Neoplasms
Keywords: OVARIAN NEOPLASMS; ADJUVANT CHEMOTHERAPY; INTRAPERITONEAL CHEMOTHERAPY
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IP Chemotherapy (Experimental): Patients with optimally debulked advanced (stage 3 or 4) epithelial ovarian cancer; IV Paclitaxel 175mg/m2 + IV Carboplatin (AUC4.5) AT DAY 1; IP Paclitaxel 60 mg/m2 at day 8; every 21 days, 6 cycles
  Interventions: Drug: IP chemotherapy

INTERVENTIONS:
Drug: IP chemotherapy — IV Paclitaxel 175mg/m2 + IV Carboplatin (AUC4.5) AT DAY 1; IP Paclitaxel 60 mg/m2 at day 8; every 21 days, 6 cycles
  Other Names: Paclitaxel; Carboplatin

SUMMARY:
Most patients with advanced ovarian cancer suffered recurrences. Therefore, adjuvant therapy is recommended for all patients with advanced ovarian cancer.

Traditionally, intravenous paclitaxel + carboplatin has been the standard adjuvant therapy.

Recently, intraperitoneal combination chemotherapy has been reported to be effective in ovarian cancer.

We attempted to evaluate the efficacy and feasibility of standard intravenous paclitaxel + carboplatin plus intraperitoneal paclitaxel chemotherapy.

DETAILED DESCRIPTION:
Epithelial ovarian cancer is the leading cause of death from gynecologic malignancies worldwide. The recommended treatment includes primary surgery for diagnosis, staging, and cytoreduction, followed by chemotherapy. Epithelial ovarian cancer is more sensitive to cytotoxic drugs than other solid tumors, most patients with advanced ovarian cancer are recommended treatment with postoperative adjuvant chemotherapy. The recommended initial chemotherapy is generally platinum and taxane combination given by intravenous infusion every 3 weeks for 6 courses. This treatment resulted in complete remission in about 50% of ovarian cancer patients and pathologic complete response in 25~30% of patients.

However most patients with advanced ovarian cancer suffered recurrences after primary treatment, median progression free survival is 15.5-22months, and median overall survival is about 31-44months.

As residual ovarian cancer after surgery and initial recurrences are primarily confined to the abdomen, intraperitoneal administration of chemotherapy was proposed several decades ago. In 2006, Armstrong, et al., reported improvement of overall survival in ovarian cancer patient with optimal surgical debulking followed intraperitoneal paclitaxel + cisplatin chemotherapy. The National Cancer Institute (NCI) of the United States recommended to consider intraperitoneal chemotherapy in optimally debulking patients.

In Korea, however, there are few studies about postoperative adjuvant intraperitoneal chemotherapy in optimally debulked (residual mass <1cm) advanced ovarian cancer patients.

Therefore the investigators tend to evaluate the efficacy and feasibility of postoperative adjuvant intraperitoneal chemotherapy. (standard intravenous paclitaxel+carboplatin plus intraperitoneal paclitaxel chemotherapy)

ELIGIBILITY:
Inclusion criteria:

1. Age >=20 and <=75
2. Histologically confirmed epithelial ovarian cancer, primary peritoneal carcinoma, tubal cancer
3. Stage 3 or 4
4. WBC >= 3500/mm3, ANC >= 1500/mm3, platelet >= 100000/mm3, hemoglobin >= 10 g/dl
5. Serum creatinine <= upper normal limit * 1.25
6. Total bilirubin <= 1.5mg/mm3, ALT/AST <= upper normal limit * 3, ALP <= upper normal limit * 3
7. Adequate compliance and geographical closeness which make adequate follow-up possible
8. GOG performance status 0-2
9. Anticipated survival >= 3 months
10. Who agreed to participate in this study and signed on informed consent form

Exclusion criteria:

1. History of chemotherapy or radiotherapy on abdomen/pelvis area
2. Pleural/pericardial effusion, ascites causing respiratory difficulties >= NCI-CTCAE grade 2
3. History of other cancers within 5 years
4. History of unapproved therapy within 30 days before enrollment
5. Other serious diseases which could threat the safety of participants or impair the ability of participants to complete the participation.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
2 year progression-free survival rate. | 2 Year after initial surgery
  The time from randomization to the time of disease progression as determined by the investigator or death from any cause.
  Progression is diagnosed by imaging or serial tumor marker elevation.

SECONDARY OUTCOMES:
Median overall survival | From entry into the study to 5 year after treatment or until half of participants are dead
  Median observed length of life from entry into the study to death; or for living patients, the date of last contact regardless of whether or not this contact is on a subsequent protocol
5 year progression-free survival rate | 5 year after initial surgery
  The time from randomization to the time of disease progression as determined by the investigator (by clinical, radiological or pathological means) or death from any cause
5 year overall survival rate | 5 year after initial surgery
  Observed length of life from entry into the study to death; or for living patients, the date of last contact regardless of whether or not this contact is on a subsequent protocol.

CONTACTS AND LOCATIONS:
Overall Officials: SANG YOUNG RYU, M.D., Principal Investigator — KOREA CANCER CENTER HOSPITAL, KOREA INSTITUTE OF RADIOLOGICAL & MEDICAL SCIENCES
Locations (1):
- Korea Cancer Center Hospital, Korea Institute of Radiological & Medical Sciences, Seoul, South Korea